CLINICAL TRIAL: NCT03297125
Title: Assessment of Optune Therapy for Patients With Newly Diagnosed Glioblastoma Using Advanced MRI
Status: Active, not recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jennifer Connelly, MD, Associate Professor, Medical College of Wisconsin
Other Study IDs: PRO00000087
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma
Keywords: Optune Therapy; MRI; NovoCure-TTF-200A
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Eligible Subjects: All enrolled subjects undergoing Optune therapy.
  Interventions: Device: Standard Magnetic Resonance Imaging (MRI); Device: Advanced MRI.

INTERVENTIONS:
Device: Standard Magnetic Resonance Imaging (MRI) — Standard MRI.
Device: Advanced MRI. — Perfusion and diffusion MRI.

SUMMARY:
The purpose of this prospective, nonrandomized controlled phase IV study is to compare standard and advanced MRI for their ability to predict response to Optune therapy.

DETAILED DESCRIPTION:
Protocol Summary: Optune therapy is a newly approved treatment for patients with glioblastoma. This therapy demonstrated comparable outcomes for patients with recurrent GBM, in comparison to standard therapies, but better quality of life. More recently, in an interim analysis of 315 patients with GBM, adding Tumor Treating Fields (TTFields) to maintenance temozolomide chemotherapy significantly prolonged progression-free and overall survival. It also has demonstrated promise in other cancers such as pancreas, mesothelioma, ovarian and lung. However, in order to optimize the treatment regimen, and potentially predict which patients are most likely to respond, reliable ways of evaluation are necessary. Advanced perfusion and diffusion MRI methods have shown utility with other treatments such as bevacizumab. Preliminary data suggests the same might be true for the evaluation of Optune therapy. The team therefore proposes to determine the utility of these methods to predict response to Optune therapy. A successful result will have wide-ranging implications not only for the optimization of Optune treatment of brain cancer but also other cancers shown to benefit from this novel therapy.

Objective: To compare standard and advanced MRI for their ability to predict response to Optune therapy. The team's approach will be to obtain both standard and advanced MRI in patients with newly diagnosed glioblastoma undergoing adjuvant chemotherapy plus Optune therapy. The ability of standard and advanced MRI to predict response will be assessed. The hypothesis is that perfusion and/or diffusion imaging metrics can be used to predict response to and elucidate mechanisms of action for Optune treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed glioblastoma (GBM), World Health Organization (WHO) grade IV.

Exclusion Criteria:

* Optune compliance < 75%; they would be excluded from the final analyses.
* History of craniectomy or significant skull defect (contraindication to Optune).
* Active implantable medical device (e.g., deep brain stimulator (DBS), spinal cord stimulator, pacemaker, defibrillator, vagus nerve stimulator, programmable shunt).
* Karnofsky Performance Status (KPS) < 60.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with newly diagnosed or recurrent glioblastoma who have self-selected Optune therapy (group 1) or declined Optune therapy (group 2).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival. | Six months.
  The number of subjects alive at six months.
Overall survival. | One year.
  The number of subjects alive at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Connelly, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No